CLINICAL TRIAL: NCT03566394
Title: Primary Prophylactic Gabapentin for Taxane-Induced Arthralgia and Myalgia Syndrome in Breast Cancer Patients Undergoing Adjuvant Chemotherapy: A Randomized Controlled Trial
Brief Title: Prophylactic Gabapentin for Taxane-Induced Arthralgia and Myalgia Syndrome in Breast Cancer Patients Undergoing Adjuvant Chemotherapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gabapentin RCT
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Invasive Breast Cancer; Chemotherapeutic Toxicity; Myalgia; Arthralgia
MeSH Terms: conditions — Myalgia; Arthralgia | interventions — Gabapentin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prophylactic Gabapentin (Experimental): Gabapentin at a dose of 300mg three times a day for 2 days before and 5 days after each taxane infusion. Administered orally.
  Interventions: Drug: Gabapentin 300mg
- Observation (No Intervention)

INTERVENTIONS:
Drug: Gabapentin 300mg — Gabapentin 300mg orally three times a day, from 2 days before to 5 days after taxane infusion
  Arms: Prophylactic Gabapentin

SUMMARY:
Taxane-induced arthralgia and myalgia syndrome (TAMS) is one of the most common side effects of taxane chemotherapy. This prospective randomized controlled trial will evaluate the efficacy of gabapentin administered prophylactically on days -2 to +5 during the taxane-portion of chemotherapy for adjuvant breast cancer patients on reducing TAMS. This will be compared to observation alone.

DETAILED DESCRIPTION:
The taxanes are a class of anticancer agents that interfere with microtubule disassembly. They have been an integral part of adjuvant breast cancer treatment since the early 2000s. Taxane-induced arthralgia and myalgia syndrome (TAMS) is one of the most common side effects of taxane chemotherapy. It is characterized by muscle and joint pain that often starts 24-48 hours after taxane-based chemotherapy, and lasts for 5-7 days. TAMS can significantly impact the level of functioning and quality of life of early-stage breast cancer patients and can occur in up to 87% of women during their chemotherapy.

Many studies have been conducted looking at medications to prevent TAMS. Unfortunately, these are primarily small retrospective or case series studies, and no standard of care has been established. Results from studies looking at antihistamines, corticosteroids, opioids, amifostine, glutamine, Shakuyaku-Kanzou-to (a Japanese herbal medicine), are conflicting and/or inconclusive.

Gabapentin, a structural analog of gamma amino butyric acid (GABA), is a second-line antiepileptic and is also widely used to treat neuropathic pain syndromes. Many oncologists already use prophylactic gabapentin in an attempt to prevent TAMS, however this is supported primarily by small case series and retrospective data, and is not considered standard of care. Unfortunately, a systemic review found no randomized controlled trial evidence supporting these findings.

This prospective randomized controlled trial will be conducted to evaluate the efficacy of gabapentin administered prophylactically on days -2 to +5 during the taxane-portion of chemotherapy for adjuvant breast cancer patients on reducing TAMS. The hypothesis for this study is that prophylactic gabapentin is more effective than observation in reducing the severity of taxane-induced arthralgias and myalgias syndrome in breast cancer patients undergoing adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Patients must have histologically confirmed, Stage I-III, breast cancer
* Patient is on an 8-cycle adjuvant anthracycline-cyclophosphamide-taxane containing chemotherapy regimen, and will be starting the taxane-containing portion of chemotherapy within 4 weeks of enrollment.
* Patient has not received prior taxane chemotherapy
* ECOG performance status 0 to 2 (on a scale from 0 to 4, with 0 indicating normal activity, 1 symptomatic but ambulatory self-care possible, 2 ambulatory more than 50% of the time, 3 ambulatory 50% of the time or less and nursing care required, and 4 bedridden and possibly requiring hospitalization)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients on FEC-D, ACTW, DCx4 chemotherapy.
* Metastatic disease
* Patient currently taking gabapentin or pregabalin for other indications prior to initiating chemotherapy
* Patients concomitantly taking other drugs known to influence GABA (e.g. barbituates, benzodiazepines, nonbenzodiazepines, baclofen)
* Patients using selected analgesics (opioids, acetaminophen, aspirin, NSAIDs) in which the dosages have changed in the 2 weeks prior to starting Taxane chemotherapy, or an analgesic medication was discontinued in the last 2 weeks, or a new analgesic medication was started in the last 2 weeks.
* Patients concomitantly using medical marijuana
* Known restricting adverse events or allergy to gabapentin or pregabalin supplements.
* GFR less than 30ml/min
* Myalgia and/or arthralgia unrelated to chemotherapy, or severe pain syndromes, that could confound the results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-07-02 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
"Worst" pain score | Approximately 8 months
  Brief Pain Inventory-short form assessment tool

SECONDARY OUTCOMES:
Arithmetic mean of the four severity pain score items | Approximately 8 months
  Brief Pain Inventory-short form assessment tool
Quality of life and function | Approximately 8 months
  FACT-Taxane Scale
Chemotherapy dose reductions, delays, and discontinuation | Approximately 8 months
Incidence and severity of peripheral neuropathy | Approximately 8 months
  EORTC-QLQ-CIPN20
Gabapentin-related adverse events | Approximately 8 months
Opioid initiation or modifications | Approximately 8 months

IPD SHARING:
Plan to Share IPD: No